CLINICAL TRIAL: NCT06494865
Title: " Role of Diffusion Weighted Image in the Diagnosis and Follow up of Breast Cancer"
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mennatallah Ashraf Ibrahim, Resident-radiology department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-24-06-23MS
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI device — Standered breast coils with small field of veiw and thin sections will be used for the examinatio.
  MRI breast including Axial T1WI, T2WI Stir contrast DWI and Stir sagittal T1WI with contrast traction and subtraction

SUMMARY:
Breast MRI has become an important tool for breast cancer detection and characterization.Contrast enhanced MRI(CE-MRI) is currently the most sensitive detection technique for diagnosis of breast cancer.

DETAILED DESCRIPTION:
Most of the lesions that occur in the breast are benign lesions. It is important to recognize benign lesions and distinguish them from breast cancer.

Nowadays sonomammography still represents the primary imaging modality utilized for breast cancer screening and diagnosis.

Breast MRI has become an important tool for breast cancer detection and characterization.Contrast enhanced MRI(CE-MRI) is currently the most sensitive detection technique for diagnosis of breast cancer.Diffusion weighted imaging provides micro-structural informations regadrding the diffusion of the water molecules in the tissue cellularity and tissue structure by using the quantitive analysis with the apparent diffusion coefficient (ADC) values.

Using Diffusion weighted imaging (DWI) combined to MRI is helpful to distinguish malignant versus benign breast lesions and it also may reduce the number of unnecessarily breast biopsies.

ELIGIBILITY:
Inclusion Criteria:

* * Female gender

  * Age more than 18 years
  * Patients presented with breast lump
  * Patients with recurrent breast cancer following chemotherapy or radiotherapy sessions.

Exclusion Criteria:

* Male gender

  * Age younger than 18 years
  * Patients with recent breast trauma in the same diseased breast within the last 6 months
  * Lactating female presented with acute symptoms as trauma or breast abscess
  * Contraindication to perform MRI examination .these include : Cardiac pacemaker -Metallic aneurysm clips

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female gender
  * Age more than 18 years
  * Patients presented with breast lump
  * Pateints with recurrent breast cancer following chemotherapy or radiotherapy sessions.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of correlated false positive results of MRI DWI for the lesion with the positive results by histopathology. | 6 months
  evaluation of the lesion with MRI DWI and histopathology for detect rate of false posive results

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stachs A, Stubert J, Reimer T, Hartmann S. Benign Breast Disease in Women. Dtsch Arztebl Int. 2019 Aug 9;116(33-34):565-574. doi: 10.3238/arztebl.2019.0565. PMID 31554551
- [Background] Butti R, Das S, Gunasekaran VP, Yadav AS, Kumar D, Kundu GC. Receptor tyrosine kinases (RTKs) in breast cancer: signaling, therapeutic implications and challenges. Mol Cancer. 2018 Feb 19;17(1):34. doi: 10.1186/s12943-018-0797-x. PMID 29455658
- [Background] Shi RY, Yao QY, Wu LM, Xu JR. Breast Lesions: Diagnosis Using Diffusion Weighted Imaging at 1.5T and 3.0T-Systematic Review and Meta-analysis. Clin Breast Cancer. 2018 Jun;18(3):e305-e320. doi: 10.1016/j.clbc.2017.06.011. Epub 2017 Jul 5. PMID 28802529
- [Background] Yilmaz E, Sari O, Yilmaz A, Ucar N, Aslan A, Inan I, Parlakkilic UT. Diffusion-Weighted Imaging for the Discrimination of Benign and Malignant Breast Masses; Utility of ADC and Relative ADC. J Belg Soc Radiol. 2018 Feb 7;102(1):24. doi: 10.5334/jbsr.1258. PMID 30039037